CLINICAL TRIAL: NCT04439162
Title: Results of Combined Antegrade and Retrograde Versurs Antegrade Cardioplegia in Complex Coronary Artery Bypass Surgeries
Brief Title: Antegrade and Retrograde Versurs Antegrade Cardioplegia in Complex Coronary Artery Bypass Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, El hussein Mohamed Abdelmotaleb Abdelhafez, associate lecteuer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: coronary artery bypass surgery
Record Dates: First submitted 2020-06-11; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Coronary Artery Disease Left Main
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group A (Experimental): antegrade cardioplegia
  Interventions: Procedure: retrograde cardioplegia protection

INTERVENTIONS:
Procedure: retrograde cardioplegia protection — antegrade-retrograde cardioplegia

SUMMARY:
During coronary artery bypass surgery, myocardial protection, especially of the right ventricle, may be inadequate in the presence of severe coronary lesions that obstruct the antegrade delivery of cold cardioplegia

DETAILED DESCRIPTION:
Asymetric myocardial cooling has been reported to yield postoperative right ventricular dysfunction, which may contribute to postoperative morbidity and mortality. Retrograde coronary sinus perfusion was introduced in 1956 to facilitate surgery involving the aortic valve. This technique was introduced as a means of myocardial protection for coronary artery bypass surgery in 1967 and has recently received renewed interest. An innovative method of delivering retrograde cardioplegia through the right atrium was recently developed by Fabiani and associates. This technique has obviated the need to directly cannulate the coronary sinus and thus has eliminated concerns regarding coronary sinus rupture due to cannulation, and concerns of inadequate right ventricular perfusion. In contrast to antegrade delivery, retrograde delivery of cardioplegia through the right atrium is not subject to the problem of limited distribution in the presence of coronary artery occlusive disease and thus allows more uniform cooling of the left ventricle,so the study will compare the results of combined antegrade and retrograde versurs antegrade cardioplegia in complex coronary artery bypass surgeries

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years
* LV ejection fraction between 30 and 50%
* left main stem CAD
* mitral or aortic valve disease associated with ischemic heart disease

Exclusion Criteria:

* Double valve disease or other valve disease
* mitral or aortic valve disease associated with congenital heart disease
* patients subjected to prior heart surgery
* emergency operation
* poorly controlled diabetes mellitus

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
myocardial function | two years
  compare simultaneous antegrade-retrograde cardioplegia with antegrade cardioplegia in coronary artery surgeries in preservation of myocardial function by using transthoracic echocardiography examination postoperatively